CLINICAL TRIAL: NCT03125265
Title: DIETary Intake, Death and Hospitalization in Adult With End-stage Kidney Disease Treated With HemoDialysis (DIET-HD) Study
Status: Completed | Type: Observational
Sponsor: Giovanni Strippoli (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Sponsor-Investigator, Giovanni Strippoli, Associate Professor, University of Bari
Organization: University of Bari (Other)
Other Study IDs: DIET-HD study
Record Dates: First submitted 2017-04-18; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Diet Habit; End Stage Renal Disease
Keywords: nutrition; hemodialysis; mortality; omega 3
MeSH Terms: conditions — Feeding Behavior; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: dietary intake of omega-3 and omega-6 polyunsaturated fatty acids

SUMMARY:
The DIETary intake, death and hospitalisation in adults with end-stage kidney disease treated with HaemoDialysis (DIET-HD) study is a multinational prospective cohort study designed to evaluate the association between nutrition and dietary patterns and health outcomes in prevalent adult haemodialysis patients in Europe and South America.

ELIGIBILITY:
Inclusion Criteria:

* End-stage kidney disease
* Long-term haemodialysis for at least the previous 90 days
* 18 years or older
* Treating team agrees to the patient's involvement in the study
* Participant willing to provide written and informed consent.-

Exclusion Criteria:

* significant neurocognitive disability or medical comorbidity that would preclude them from understanding the dietary questionnaire even if assisted
* a life expectancy less than 6 months according to their treating physician
* planned kidney transplantation within 6 months of baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: dialysis clinics administered by a single dialysis provider
Sampling Method: Non-Probability Sample
Enrollment: 9757 (Actual)
Dates: Start 2014-01-05 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Cardiovascular mortality | 12 months since baseline dietary evaluation
  Defined as sudden death or death attributed to acute myocardial infarction, pericarditis, atherosclerotic heart disease, cardiomyopathy, cardiac arrhythmia, cardiac arrest, valvular heart disease, pulmonary edema, or congestive cardiac failure

SECONDARY OUTCOMES:
All-cause mortality | 12 months since baseline dietary evaluation
Infection-related mortality | 12 months since baseline dietary evaluation
All-cause and cardiovascular related hospitalisation | 12 months since baseline dietary evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni FM Strippoli, MD, PhD — University of Bari

REFERENCES:
- Available data/document: Study Protocol — http://bmjopen.bmj.com/content/5/3/e006897.long